CLINICAL TRIAL: NCT04520945
Title: Phase 2B: Randomized Double-Blinded Clinical Study of Chondrogen for Treatment of Knee Osteoarthritis
Brief Title: Phase 2B Clinical Study of Chondrogen for Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meluha Life Sciences SDN BHD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chondrogen
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 100 patients will be selected from 2 different study sites. Each study site comprises 50 patients.
Who Masked: Participant, Investigator
Masking Description: The outcomes assessor will help to screen the participants and send them to the clinical investigators for further medical screening. The participant's personal details will be private and confidential to the outcomes assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Participant of Phase 2B Clinical Study Chondrogen (Active Comparator): 50 participants will receive the investigational drug (Chondrogen and Hyaluronic Acid) through the intra-articular injection method. The participants will receive the investigational drug one time. The injection will be provided to the participant on the baseline day.
  Interventions: Biological: Chondrogen
- Placebo Participant of Phase 2B Clinical Study Chondrogen (Placebo Comparator): 50 participants will receive the placebo (Saline and Hyaluronic Acid) through the intra-articular injection method. The participants will receive the investigational drug one time. The injection will be provided to the participant on the baseline day.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Chondrogen — Mesenchymal stem cell-derived from umbilical cord Wharton Jelly and hyaluronic acid
  Other Names: Mesenchymal Stem Cell
  Arms: Active Participant of Phase 2B Clinical Study Chondrogen
Biological: Placebo — Consist of saline and hyaluronic acid
  Arms: Placebo Participant of Phase 2B Clinical Study Chondrogen

SUMMARY:
Primary osteoarthritis is a debilitating disease characterized by extensive damage to the joints and excruciating pain leading to loss of activity and depression. Despite advances in diagnosis, the quest for the development of a disease-modifying osteoarthritis drug has proven unsuccessful. Human cartilage only has limited regenerative potential. Transplantation is a promising strategy given the high proliferative capacity of MSCs and their potential to differentiate into cartilage-producing cells - chondrocytes. The acquisition of MSC does not require invasive surgical intervention or cartilage extraction from other sites as required by other cell-based strategies. The investigators inject allogeneic human mesenchymal stem cells to the cartilage lesions in patients via intra-articular injection method, and to investigate the efficacy and safety.

DETAILED DESCRIPTION:
Osteoarthritis is one of the commonest diseases in the world, with a global disease burden of 83%. Plain radiograph remained the main modality in diagnosing osteoarthritis. Chondrogen is a mesenchymal stem cell-derived from umbilical cord tissue product. The mesenchymal stem cell is used for the study because of its ability to proliferate and differentiate into various tissues such as chondrocytes, adipocytes, and osteocytes. Various clinical studies have been conducted for arthritis, orthopedic, joint, and cartilage.

This study will enroll 100 patients age 30-70 years old. They will be divided into 2 groups which are the group which will receive the investigational drug (ChondrogenTM and HA) and another group will receive a placebo (saline and HA). It will be a randomized double-blinded study where the participants and the investigator would not know what are the things being received. This study will be conducted for 24 months. The injection will be given on the baseline day after screening the volunteers. The patients will be assessed on VAS, WOMAC, IKDC, KOOS PROMIS29, the interleukins, and MRI.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years old
* No serious infection, chronic diseases, diabetes and tuberculosis
* Idiopathic or secondary osteoarthritis of the knee with grade 1-3 defined by the modified Kellgren-lawrence classification
* Written informed consents were obtained from all subjects.

Exclusion Criteria:

* Pregnant or lactating women
* Women of childbearing potential unwilling to use two forms of contraception
* Cognitively impaired adults
* Presence of large meniscal tears
* Inflammatory or post-infectious arthritis
* More than 5 degrees of varus or valgus deformity
* Kellgren Lawrence grade 4 osteoarthritis in two compartments in persons over 60 years of age
* Intra-articular corticosteroid injection within the 3 previous months
* Major neurologic deficit
* Arthroscopy during the previous 6 months
* Poorly controlled diabetes mellitus
* Immunosuppressive or anticoagulant treatment
* NSAID therapy within 15 days prior to inclusion in the study
* Serious medical illness with a life expectancy of less than 1 year
* Prior admission for substance abuse
* Body Mass Index (BMI) of 40 kg/m2 or greater
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
VAS score | 12 months
  Change from Baseline in Visual Analogue Scale (VAS)
WOMAC score | 12 months
  Change from Baseline in Western Ontario and McMaster Universities Osteoarthritis Index Score (WOMAC)
IKDC score | 12 months
  Change from Baseline in knee function change and improvement (IKDC)
KOOS score | 12 months
  Change from Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS)

SECONDARY OUTCOMES:
PROMIS29 score | 12 months
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS29) scores
Kellegren-Lawrence grading | 12 months
  Number of participants evaluated by X-ray and MRI of knee OA from baseline Kellegren-Lawrence grading system.
Interleukins | 12 months
  Changes of interleukins (IL-1b, IL-6, PGE-2, TGF-b, TNF-a, IGF-1) of articular cavity fluid from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Badrul Akmal Hisham, MBBS, Principal Investigator — PPUKM
Locations (1):
- Department of Orthopedic & Traumatology, Faculty of Medicine, Hospital Canselor Tuanku Mukhriz, UKM Medical Centre, Jalan Yaacob Latiff, Bandar Tun Razak, Cheras, 56000 Kuala Lumpur., Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No